CLINICAL TRIAL: NCT04767490
Title: Single Anastomosis Versus Standard Duodenal Switch - a Prospective Randomized Single-blinded Trial
Brief Title: Single Anastomosis Versus Standard Duodenal Switch
Acronym: SADI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Institut universitaire de cardiologie et de pneumologie de Québec, University Laval (Other)
Responsible Party: Principal Investigator, Laurent Biertho, Principal Investigator, Laval University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SADI
Record Dates: First submitted 2018-03-23; First posted 2021-02-23 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Obesity; Morbid Obesity
Keywords: bariatric surgery
MeSH Terms: conditions — Obesity; Obesity, Morbid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BPD-DS (Active Comparator): Biliopancreatic diversion with Duodenal Switch (BPD-DS), with Sleeve gastrectomy, including a 100cm common channel and 150cm stric alimentary limb
  Interventions: Procedure: Standard Duodenal Switch
- SADI (Experimental): Single-Anastomosis Duodeno-Ileal anastomosis (SADI) with Sleeve Gastrectomy, including a 250cm common channel
  Interventions: Procedure: Single Anastomosis Duodenal Switch

INTERVENTIONS:
Procedure: Standard Duodenal Switch
  Other Names: BPD-DS
  Arms: BPD-DS
Procedure: Single Anastomosis Duodenal Switch
  Other Names: SADI
  Arms: SADI

SUMMARY:
Bilio-Pancreatic diversion with Duodenal Switch (BPD-DS) is the most effective bariatric procedure in terms of long-term weight loss and remission rate of Type 2 Diabetes. However, its technical difficulty and increased risk of long-term nutritional deficiencies have been a major hindrance to its diffusion.

Recently, a " simplified " technique of Duodenal-Switch has been proposed by Sanchez-Pernaute et al. This technique involves the creation of a Sleeve Gastrectomy, transection of the first duodenum, and connection of the duodenum to an omega-loop of small bowel instead of a terminal intestinal loop used in standard BPD-DS.

The overall objective of this study is to assess in a prospective randomized blinded trial, the outcomes of this new procedure, using a comprehensive clinical evaluation and follow-up method. This could potentially change the clinical practice and surgical approach in our Institution.

DETAILED DESCRIPTION:
Bilio-Pancreatic diversion with Duodenal Switch (BPD-DS) is the most effective bariatric procedure in terms of long-term weight loss and remission rate of Type 2 Diabetes. However, its technical difficulty and increased risk of long-term nutritional deficiencies have been a major hindrance to its diffusion. Our team, with more than 4000 BPD-DS performed since the early 1990's, is recognized internationally for its expertise with this specific procedure.

Recently, a " simplified " technique of Duodenal-Switch has been proposed by Sanchez-Pernaute et al. This technique involves the creation of a Sleeve Gastrectomy, transection of the first duodenum, and connection of the duodenum to an omega-loop of small bowel instead of a terminal intestinal loop used in standard BPD-DS.

This new procedure, called Single Anastomosis Duodenal Switch has the potential benefit of decreasing the complexity of the standard BPD-DS by avoiding one of the two intestinal anastomoses usually needed. This could potentially decrease the rate of peri-operative complications and increase access to this type of surgery.

However, the length of the common channel (250cm) is more than doubled compared to standard BPD-DS, which could also change significantly the outcomes of the procedure itself. Indeed, the length of the common channel conditions the absorption of fat and fat-soluble vitamins.

Currently, the scientific literature regarding this procedure is scarce, with only one author who published his 2-years outcomes, in a cohort study of 100 patients. In addition, this report presents major limitations. In example, the length of the omega loop was increased from 200 to 250cm during the course of the study, in order to decrease the rate of protein deficiency and reoperation for malnutrition. This and other limitations make it hard to assess the actual results of the technique.

The overall objective of this study is to assess in a stronger study design (i.e. a prospective randomized single blinded trial), the outcomes of this new procedure, using a comprehensive clinical evaluation and follow-up method. This could potentially change the clinical practice and surgical approach in our Institution.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years and ≤60 years
* Fulfill criteria for bariatric surgery as coined by National Institutes of Health BMI≥35
* Give written informed consent

Exclusion Criteria:

Participants who meet any of the following criteria at the time of the baseline visit are excluded from the study:

* Presence of the following baseline comorbidities:
* Inflammatory bowel disease (IBD),
* Cirrhosis
* History of gastric or duodenal ulcers
* Preoperative hypoalbuminemia (<35 g/L)
* History of severe renal, hepatic, cardiac or pulmonary disease
* Past esophageal, gastric or bariatric surgery
* Type 1 Diabetes
* Pregnancy
* Evidence of psychological problem that may affect the capacity to understand the project and to comply with the medical recommendations
* History of drug use or alcohol abuse in the last 6 months
* History of gastro-intestinal inflammatory diseases

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-09-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Excess weight loss | 2 years
  Excess weight loss at 2 years of follow-up
  %EWL (Excess weight loss based on an ideal BMI = 25.) and change in BMI as compared to preoperative reference values
Rate of protein deficiency or insufficiency | from baseline up to 60 months
  Rate of protein deficiency (<35gr/l) or insufficiency (<30gr/l)
Mortality rate | from baseline up to 60 months
  Rate of mortality
BMI | 2 years
  change in BMI at 2 years follow-up as compared to preoperative reference values

SECONDARY OUTCOMES:
Complication rate | from baseline up to 60 months
  overall and surgery-specific complications
Cure rate of comorbidities | from baseline up to 60 months
  Remission rate for comorbidities, including T2D, Hypertension, dyslipidemia, sleep apnea
Rate of minerals and vitamin deficiencies | from baseline up to 60 months
  Rate of deficiency and insufficiency in mineral and vitamins
Body composition by bioimpedance measures | from baseline up to 60 months
  body fat composition (%) assessed by biompedance
Change in quality of life | from baseline up to 60 months
  36-item short form survey score from 0 to 100
Change in quality of life | from baseline up to 60 months
  Bariatric Analysis and Reporting Outcomes System score from -7 to 9
Change in quality of life | from baseline up to 60 months
  Laval Questionnaire score from 0 to 7
Change in quality of life | from baseline up to 60 months
  GastroIntestinal Quality of Life Index from 0 to 144
Change in gatroesophageal reflux symptom | from baseline to 60 months
  GastroEsophageal Reflus Disease Score from 0 to 72

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Biertho, MD, Principal Investigator — Institut universitaire de cardiologie et de pneumologie de Québec, University Laval
Locations (1):
- Institut Universitaire de Cardiologie et de Pneumologie de Québec, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No